CLINICAL TRIAL: NCT03572933
Title: A Double-blind, Randomized, Placebo-controlled Trial of Adjunctive Ganaxolone Treatment in Children and Young Adults With Cyclin-dependent Kinase-like 5 (CDKL5) Deficiency Disorder (CDD) Followed by Long-term Open-label Treatment
Brief Title: Study of Adjunctive Ganaxolone Treatment in Children and Young Adults With CDKL5 Deficiency Disorder
Acronym: Marigold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-CDD-3001; 2018-001180-23 (EudraCT Number)
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: CDKL5 Deficiency Disorder
Keywords: refractory seizures; genetic pediatric encephalopathies; epilepsy in children; seizure disorder
MeSH Terms: conditions — CDKL5 deficiency disorder; Seizures; Epilepsy | interventions — ganaxolone

STUDY DESIGN:
Intervention Model Description: The double-blind phase will randomize subjects to adjunctive ganaxolone or placebo at a 1:1 ratio to standard of care
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ganaxolone (Experimental): ganaxolone suspension (50 mg/ml) 3x's /day for 17 weeks
  Interventions: Drug: ganaxolone
- Placebo (Placebo Comparator): placebo suspension 3x's /day for 17 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ganaxolone — active drug
  Arms: Ganaxolone
Drug: Placebo — inactive
  Other Names: Placebo (for ganaxolone)
  Arms: Placebo

SUMMARY:
A clinical study to evaluate the efficacy, safety, and tolerability of adjunctive ganaxolone therapy compared to placebo for the treatment of seizures in children and young adults with genetically confirmed CDKL5 gene mutation.

DETAILED DESCRIPTION:
The Marigold Study is a global, double-blind, placebo-controlled, Phase 3 clinical trial that will enroll approximately 70 patients between the ages of 2 and 21 with a confirmed disease-related CDKL5 gene variant. Patients will undergo a baseline period before being randomized to receive, in addition to their existing anti-seizure treatment, either ganaxolone or placebo for 17 weeks. Following the treatment period, all patients that meet certain eligibility requirements will have the opportunity to receive ganaxolone in the open label phase of the study. The study's primary efficacy endpoint is percent reduction in seizures. Secondary outcome measures will include non-seizure-related endpoints to capture certain behavioral and sleep disturbances that have been seen in previous clinical studies with ganaxolone.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed CDKL5 gene mutation, seizure onset by 1 year of age and lack of independent ambulation by 2 years of age
* Failure to control seizures despite 2 or more anti-seizure medications
* At least 16 seizures per 28 days of primary seizure types
* On a stable regimen of 0-4 anti-seizure medications (Vagus nerve stimulator, ketogenic diet, and modified Atkins diet do not count towards this limit)
* Additional Inclusion Criteria apply and can be discussed with study team

Exclusion Criteria:

* Previous exposure to ganaxolone
* West Syndrome with hypsarrhythmia pattern on EEG or seizures predominantly of Infantile Spasms type
* Use of adrenocorticotropic hormone (ACTH), prednisone or other glucocorticoid or use of moderate or strong inducers or inhibitors of CYP3A4/5/7 are prohibited
* Use of tetrahydrocannabinol (THC) or cannabidiol (CBD) is prohibited during the double-blind phase, unless patient has a prescription of Epidiolex®
* Exposure to any other investigational drug within 30 days or fewer than 5 half-lives prior to screening
* Plasma allopregnanolone-sulfate (Allo-S) levels greater than or equal to 6.0 ng/ml at screening visit
* Additional Exclusion Criteria apply and can be discussed with study team

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hulihan, MD, Study Director — Marinus Pharmaceuticals, Inc.
Locations (36):
- United States (17):
  - Marinus Research Site, Phoenix, Arizona
  - Marinus Research Site, Los Angeles, California
  - Marinus Research Site, Aurora, Colorado
  - Marinus Research Site, Gulf Breeze, Florida
  - Marinus Research Site, Orlando, Florida
  - Marinus Research Site, Norcross, Georgia
  - Marinus Research Site, Chicago, Illinois
  - Marinus Research Site, Iowa City, Iowa
  - Marinus Research Site, Boston, Massachusetts
  - Marinus Research Site, Rochester, Minnesota
  - Marinus Research Site, St Louis, Missouri
  - Marinus Research Site, Livingston, New Jersey
  - Marinus Research Site, Cleveland, Ohio
  - Marinus Research Site, Philadelphia, Pennsylvania
  - Marinus Research Site, Pittsburgh, Pennsylvania
  - Marinus Research Site, Fort Worth, Texas
  - Marinus Research Site, Houston, Texas
- Australia (3):
  - Marinus Research Site, Brisbane, Queensland
  - Marinus Research Site, Heidelberg, Victoria
  - Marinus Research Site, Melbourne, Victoria
- Marinus Research Site, Paris, France
- Marinus Research Site, Ramat Gan, Israel
- Italy (5):
  - Marinus Research Site, Florence
  - Marinus Research Site, Milan
  - Marinus Research Site, Pavia
  - Marinus Research Site, Roma
  - Marinus Research Site, Verona
- Poland (2):
  - Marinus Research Site, Bydgoszcz
  - Marinus Research Site, Krakow
- Russia (3):
  - Marinus Research Site, Moscow
  - Marinus Research Site, Nizhny Novgorod
  - Marinus Research Site, Novosibirsk
- United Kingdom (4):
  - Marinus Research Site, Birmingham
  - Marinus Research Site, Bristol
  - Marinus Research Facility, Glasgow
  - Marinus Research Site, London

REFERENCES:
- [Derived] Yasmen N, Sluter MN, Yu Y, Jiang J. Ganaxolone for management of seizures associated with CDKL5 deficiency disorder. Trends Pharmacol Sci. 2023 Feb;44(2):128-129. doi: 10.1016/j.tips.2022.11.007. Epub 2022 Dec 12. No abstract available. PMID 36517284
- [Derived] Knight EMP, Amin S, Bahi-Buisson N, Benke TA, Cross JH, Demarest ST, Olson HE, Specchio N, Fleming TR, Aimetti AA, Gasior M, Devinsky O; Marigold Trial Group. Safety and efficacy of ganaxolone in patients with CDKL5 deficiency disorder: results from the double-blind phase of a randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2022 May;21(5):417-427. doi: 10.1016/S1474-4422(22)00077-1. PMID 35429480

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ganaxolone
Started | 51 | 50
Completed | 47 | 48
Not Completed | 4 | 2
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ganaxolone | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.73 (4.382) | 6.78 (4.705) | 7.26 (4.547)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 43 | 44 | 87
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 47 | 46 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 18 | 42
  Poland | 5 | 5 | 10
  Italy | 6 | 9 | 15
  United Kingdom | 3 | 4 | 7
  Israel | 1 | 0 | 1
  Australia | 2 | 4 | 6
  France | 3 | 3 | 6
  Russia | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Summary of 28-day Seizure Frequency for Major Motor Seizure Types
Description: Summary of 28-day seizure frequency for Major Motor Seizure Types during the double-blind treatment period relative to the 6-week prospective baseline period
  Note: Summaries are based on the sum of the individual seizures, the countable seizures, and the clusters with uncountable seizures (each cluster with uncountable seizures counts as 1 seizure). Within the baseline and post baseline intervals, 28-day seizure frequency was calculated as the total number of seizures in the interval divided by the number of days with available seizure data in the interval, multiplied by 28.
Time Frame: End of the double-blind 17 week treatment period
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Seizures per day
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 51 | 49
Seizures per day
  Baseline (Median) | 49.17 [32.20 to 60.67] | 54.00 [38.24 to 106.67]
  17 week-post baseline phase (Median) | 55.50 [35.75 to 80.14] | 45.03 [31.83 to 76.03]

2. Secondary Outcome: Caregiver Global Impression of Change in Attention
Description: Caregiver global impression of change in attention during the double-blind treatment period of ganaxolone compared to placebo. Investigators and caregivers reported improvements in attention, mood, behavior and sleep via investigator narratives
Time Frame: End of the double-blind 17 week treatment period
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 51 | 50
Participants
  Very Much Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Very Much Improved - Visit 5 (End of Week 17) | 1 | 1
  Much Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Much Improved - Visit 5 (End of Week 17) | 7 | 2
  Minimally Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Minimally Improved - Visit 5 (End of Week 17) | 14 | 21
  No Change - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  No Change - Visit 5 (End of Week 17) | 23 | 18
  Minimally Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Minimally Worse - Visit 5 (End of Week 17) | 1 | 1
  Much Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Much Worse - Visit 5 (End of Week 17) | 1 | 1
  Very Much Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Very Much Worse - Visit 5 (End of Week 17) | 0 | 1

3. Secondary Outcome: Caregiver Global Impression of Change in Target Behavior
Description: Caregiver global impression of change in target behavior during the double-blind treatment period of ganaxolone compared to placebo. Investigators and caregivers reported improvements in attention, mood, behavior and sleep via investigator narratives.
Time Frame: End of the double-blind 17 week treatment period
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 51 | 50
Participants
  Very Much Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 46 | 45
  Very Much Improved - Visit 5 (End of Week 17) | 0 | 0
  Much Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 46 | 45
  Much Improved - Visit 5 (End of Week 17) | 6 | 4
  Minimally Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 46 | 45
  Minimally Improved - Visit 5 (End of Week 17) | 14 | 20
  No Change - Visit 5 (End of Week 17): number analyzed (Participants) | 46 | 45
  No Change - Visit 5 (End of Week 17) | 22 | 19
  Minimally Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 46 | 45
  Minimally Worse - Visit 5 (End of Week 17) | 1 | 2
  Much Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 46 | 45
  Much Worse - Visit 5 (End of Week 17) | 2 | 0
  Very Much Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 46 | 45
  Very Much Worse - Visit 5 (End of Week 17) | 1 | 0

4. Secondary Outcome: Clinical Global Impression of Improvement - Parent/Caregiver
Description: Clinical global impression of improvement during the double-blind treatment period of ganaxolone compared to placebo. The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses.
Time Frame: End of the double-blind 17 week treatment period
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 48 | 48
Participants
  Very Much Improved - Visit 5 (End of Week 17) - Parent/Caregiver | 1 | 0
  Much Improved - Visit 5 (End of Week 17) - Parent/Caregiver | 7 | 13
  Minimally Improved - Visit 5 (End of Week 17) - Parent/Caregiver | 13 | 17
  No Change - Visit 5 (End of Week 17) - Parent/Caregiver | 22 | 14
  Minimally Worse - Visit 5 (End of Week 17) - Parent/Caregiver | 4 | 2
  Much Worse - Visit 5 (End of Week 17) - Parent/Caregiver | 1 | 2
  Very Much Worse - Visit 5 (End of Week 17) - Parent/Caregiver | 0 | 0

5. Secondary Outcome: Clinical Global Impression of Improvement - Clinician
Description: Clinical global impression of improvement during the double-blind treatment period of ganaxolone compared to placebo
Time Frame: [Time Frame: End of the double-blind 17 week treatment period]
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 48 | 48
Participants
  Very Much Improved - Visit 5 (End of Week 17) - Clinician | 0 | 0
  Much Improved - Visit 5 (End of Week 17) - Clinician | 7 | 7
  Minimally Improved - Visit 5 (End of Week 17) - Clinician | 13 | 19
  No Change - Visit 5 (End of Week 17) - Clinician | 19 | 16
  Minimally Worse - Visit 5 (End of Week 17) - Clinician | 9 | 2
  Much Worse - Visit 5 (End of Week 17) - Clinician | 0 | 3
  Very Much Worse - Visit 5 (End of Week 17) - Clinician | 0 | 1

6. Secondary Outcome: Percentage of Seizure-free Days for Major Motor Seizure Types
Description: Percentage of Seizure-free Days for Major Motor Seizure types during the double-blind treatment period of ganaxolone compared to placebo. The major motor seizure types include bilateral tonic (sustained motor activity = 3 seconds), generalized tonic-clonic, atonic/drop, bilateral clonic, and focal to bilateral tonic-clonic.
Time Frame: End of the double-blind 17 week treatment period
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent of seizure-free days
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 51 | 50
percent of seizure-free days
  Baseline: number analyzed (Participants) | 51 | 49
  Baseline | 30.32 (27.070) | 22.57 (25.761)
  17-week-Post-Baseline Phase | 36.17 (30.932) | 32.29 (30.615)
  Arithmetic Change from Baseline: number analyzed (Participants) | 51 | 49
  Arithmetic Change from Baseline | 5.86 (15.350) | 9.62 (21.364)

7. Secondary Outcome: Arithmetic Change in Longest Seizure Free Interval, Based on Primary Seizure Types
Description: Arithmetic change in longest seizure free interval, based on primary seizure types during the double-blind treatment period of ganaxolone compared to placebo
Time Frame: End of the double-blind 17 week treatment period
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 51 | 49
days | -4.63 (14.867) | -0.02 (9.376)

8. Secondary Outcome: Caregiver Global Impression of Change in Seizure Intensity and Duration
Description: Caregiver global impression of change in seizure intensity and duration during the double-blind treatment period of ganaxolone compared to placebo. CGI-C is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.
Time Frame: End of the double-blind 17 week treatment period
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 51 | 50
Participants
  Very Much Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Very Much Improved - Visit 5 (End of Week 17) | 1 | 2
  Much Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Much Improved - Visit 5 (End of Week 17) | 5 | 15
  Minimally Improved - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Minimally Improved - Visit 5 (End of Week 17) | 11 | 11
  No Change - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  No Change - Visit 5 (End of Week 17) | 21 | 10
  4Minimally Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  4Minimally Worse - Visit 5 (End of Week 17) | 5 | 3
  Much Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Much Worse - Visit 5 (End of Week 17) | 4 | 2
  Very Much Worse - Visit 5 (End of Week 17): number analyzed (Participants) | 47 | 45
  Very Much Worse - Visit 5 (End of Week 17) | 0 | 2

ADVERSE EVENTS:
Time Frame: Screening through 17-week Double-blind Phase
Arm/Group | Placebo | Ganaxolone
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 5/51 | 6/50
Other Adverse Events (participants affected / at risk) | 45/51 | 43/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | Ganaxolone (N=50)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 1 (1)
Food Refusal (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to Stimuli (Nervous system disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=51) | Ganaxolone (N=50)
Somnolence (Nervous system disorders) | 8 (8) | 18 (20)
Seizure (Nervous system disorders) | 9 (12) | 7 (8)
Sedation (Nervous system disorders) | 2 (2) | 3 (3)
Hypersomnia (Nervous system disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2) | 2 (2)
Hyperaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 5 (6)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Ear Infection (Infections and infestations) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 4 (5) | 2 (4)
Respiratory Tract Infection Viral (Infections and infestations) | 3 (3) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 1 (2)
Nasopharyngitis (Infections and infestations) | 5 (5) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Varicella (Infections and infestations) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (12) | 5 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 4 (5) | 9 (10)
Gait Disturbance (General disorders) | 1 (1) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Insomnia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Irritability (Psychiatric disorders) | 2 (2) | 2 (2)
Body Temperature Increased (Investigations) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the study is part of a multicenter study, the first publication of the study results shall be made by the sponsor in conjunction with the sponsor's presentation of a joint, multicenter publication of the compiled and analyzed study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03572933/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT03572933/SAP_003.pdf